CLINICAL TRIAL: NCT00582608
Title: Tumor Detection Using Iodine-131-Labeled Monoclonal Antibody 8H9
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00-066
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: CNS Cancer; Neuroblastoma; Sarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Sarcoma

ARMS (1):
- 131I-8H9 and 8H9 (Experimental): This is an open-label single arm study of 131 I-8H9. injected intravenously at 10mCi/1.73m^2 dose [intended specific activity of '20mCi/mg protein] preceded by administration of 50mg/1.73m2 of unlabeled -8H9.
  Interventions: Drug: 131I-8H9; Drug: 8H9

INTERVENTIONS:
Drug: 131I-8H9 — This is an open-label single arm study of 131I-8H9, injected intravenously at 10 mCi/1.73 m^2 dose [intended specific activity of ~20 mCi/mg protein]
Drug: 8H9 — administration of 50mg/1.73m^2 of unlabeled 8H9.

SUMMARY:
The purpose of this study is to find out whether the monoclonal antibody 8H9 is useful in finding tumors in your body. Antibodies are protein found naturally in blood. They can fasten themselves to bacteria and viruses. They can stimulate white cells and blood proteins to kill tumors. The antibody 8H9 was made from mouse white cells. The white cells that secrete this antibody have been made to live for ever. They manufacture large amounts of 8H9 for patient use. Although other monoclonal antibodies have been safely tested in people, the antibody 8H9 has never been given to a human patient.

DETAILED DESCRIPTION:
To test if intravenous injections of iodine-131 labeled murine monoclonal antibody 8H9 can detect primary and metastatic solid tumors. A total of 60 patients will be accrued over a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pediatric/adolescent solid tumor (including neuroblastoma, rhabdomyosarcoma, Ewing's/PNET, osteosarcoma, brain tumors, desmoplastic small round cell tumor (DSRT) and other tumors that are 8H9-positive) confirmed by the MSKCC Department of Pathology.
* Patient must have either recurrent disease or have <20% chance of long term disease-free survival.
* Patient must be at least 1 year old. Age can range from 1-50 years of age.
* Patients should have measurable or evaluable disease. For tumor types that are known to be 8H9-positive, patients can be imaged after the diagnosis is made, prior to definitive surgery or surgery to confirm tumor recurrence.
* Tumor tissue is or will be available for 8H9 immunostaining. For patients with tumor-types known to be 8H9-positive, surgical samples obtained after 131I- 8H9 imaging will be immunostained to confirm 8H9-reactivity. These tumor types include: neuroblastoma, rhabdomyosarcoma, osteosarcoma, DSRT, Ewing's Sarcoma/PNET), brain tumors (glioblastoma multiforme, mixed glioma, astrocytoma, ependymoma, medulloblastoma, schwannoma., meningioma).
* If frozen tumor tissue is unavailable, and if bone marrow involvement is demonstrated by histology, 8H9 immunostaining by immunofluorescence will be carried out on patient's bone marrow. In this case, patients will be eligible for study if bone marrow 8H9 immunostaining is positive.

Exclusion Criteria:

* Severe major organ toxicity. Specifically, renal, cardiac, hepatic, pulmonary, gastrointestinal, and neurologic system toxicity should all be less than grade 2. Patients with stable neurological deficits (because of their brain tumor) are not excluded. Patients with <= 3 hearing loss are not excluded.
* Clinically apparent infections.
* History of allergy to iodine or mouse proteins.
* Patients previously treated with mouse monoclonal antibodies are not eligible unless they have no circulating HAMA.
* Pregnant women are excluded for fear of danger to the fetus. Therefore negative pregnancy test is required for all women of child-bearing age, and appropriate contraception is used during the study period.
* Patient's own tumor is negative by 8H9 immunostaining.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2001-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- MAB 131-I LABELED 8H9: MAB 131-I LABELED 8H9: This is an open-label single arm study of 131I-8H9, injected intravenously at 10 mCi/1.73 m2 dose [intended specific activity of ~20 mCi/mg protein] preceded by administration of 50mg/1.73m2 of unlabeled 8H9.
Period: Overall Study
Arm/Group | MAB 131-I LABELED 8H9
Started | 12
Completed | 0
Not Completed | 12
Not completed — Not Treated | 7
Not completed — Patient Ineligible | 1
Not completed — Lack of accrual | 4

BASELINE CHARACTERISTICS:
Arm/Group | MAB 131-I LABELED 8H9
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 7
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety and Toxicity is Measured by the Total Number of Participants Affected
Description: Safety and toxicity is measured by the total number of participants affected. Please see the adverse event table for the specifics for this protocol.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | MAB 131-I LABELED 8H9
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Arm/Group | MAB 131-I LABELED 8H9
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAB 131-I LABELED 8H9 (N=5)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAB 131-I LABELED 8H9 (N=5)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (4)
Leukocyte count decreased (Blood and lymphatic system disorders) | 2 (2)
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 (3)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Serum calcium decreased (Blood and lymphatic system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Technical problems led to unreliable and uninterpretable data. Therefore, there is no data to report under Outcome Measures. Due to lack of patients accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes